CLINICAL TRIAL: NCT03716089
Title: Prospective Controlled Clinical Trial for Comparison of Tumor Efficacy Safety in Laparoscopic Resection of Gastrointestinal Stromal Tumors Between Favorable and Unfavorable Site（FUGES-016）
Brief Title: Comparison of Tumor Efficacy Safety in Laparoscopic Resection of Gastrointestinal Stromal Tumors Between Favorable and Unfavorable Site
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Other Study IDs: FUGES-016
Record Dates: First submitted 2018-10-14; First posted 2018-10-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: GIST of Stomach; Gastric Cancer; Surgery; Complication
Keywords: GIST; laparoscopic resection; early complication; mortality; tumor sites
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (Study group): Group for laparoscopic resection of GIST with unfavorable group (Unfavorable group)
  Interventions: Procedure: Laparoscopic resection
- Group B (Control group): Group for laparoscopic resection of GIST with favorable group (favorable group)
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Laparoscopic resection — Laparoscopic surgery under general anesthesia

SUMMARY:
Participants with gastrointestinal stromal tumors(GIST) were divided into favorable and unfavorable sites according to the anatomical site of the tumor, and this study aims to validate the overall postoperative morbidity and mortality rates between favorable site receiving laparoscopic resection of GIST and that of unfavorable site under the currently standard surgical therapy.

DETAILED DESCRIPTION:
Participants with gastrointestinal stromal tumors(GIST) were divided into favorable and unfavorable sites according to the anatomical site of the tumor, and this study aims to validate the overall postoperative morbidity and mortality rates between favorable site receiving laparoscopic resection of GIST and that of unfavorable site under the currently standard surgical therapy. Main end of study: 3-year disease free survival rate

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old
2. Primary gastric lesion confirmed pathologically GIST by endoscopic biopsy. Preoperative endoscopy, ultrasound endoscopy or computer tomography, Magnetic resonance suspected GIST, and then postoperative pathology confirmed as the original GIST
3. Written informed consent
4. Expected R0 resection by laparoscopy
5. Performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) class I to III
7. Maximum tumor diameter ≤10cm

Exclusion Criteria:

1. Pregnant and lactating women
2. Suffering from a severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
4. History of previous gastric surgery (including ESD/EMR for gastric cancer)
5. Rejection of laparoscopic resection
6. History of other malignant disease within the past five years
7. History of unstable angina or myocardial infarction within the past six months
8. History of a cerebrovascular accident within the past six months
9. History of continuous systematic administration of corticosteroids within one month
10. Requirement of simultaneous surgery for another disease
11. Emergency surgery due to complications (bleeding, obstruction or perforation) caused by gastric cancer
12. FEV1<50% of the predicted values
13. Maximum tumor diameter >10cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion criteria and not conform to the exclusion criteria are qualified for this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months
  Definition of recurrence and recurrence date The following situations are regarded as "recurrence"
  1. Recurrence identified by any one image examination (X-ray, ultrasound, computed tomography, magnetic resonance imaging, etc.) and, if there are a variety of imaging examinations, results without contradiction determined "recurrence". The earliest date that the recurrence is found is defined as the "recurrence date".
  2. For cases that lack the use of imaging or a pathological diagnosis, the date of diagnosing the occurrence of clinical recurrence based on clinical history and physical examination is defined as the "recurrence date".
  3. For cases without imaging or clinical diagnosis but with a cytology or tissue biopsy pathological diagnosis of recurrence, the earliest date confirmed by cytology or biopsy pathology is considered the "recurrence date".
  4. A rise in carcinoembryonic antigen or other associated tumor markers alone could not be diagnosed as a relapse.

SECONDARY OUTCOMES:
Intraoperative morbidity rates | 30 days
  1. . The number of all patients treated with surgery as the denominator and the number of the patients with any intraoperative morbidity as the numerator are used to calculate the proportions.
  2. . Intraoperative morbidity (occurring from skin incision to skin closure) including: surgery-related morbidity: intraoperative hemorrhage and injury:
Conversion to open surgery rate | 30 days
  1. . In this study, if the length of the auxiliary incision is more than 10 cm, it is considered a conversion to open surgery.
  2. .The number of all patients treated with surgery as the denominator and the number of the patients with conversion to open surgery as the numerator are used to calculate the proportions.
Positive surgical margin rate | 30 days
  1. . The investigators confirm the surgical margin status by postoperative pathology report.
  2. . The number of all patients treated with surgery as the denominator and the number of the patients with positive surgical margin as the numerator are used to calculate the proportions.
Overall postoperative serious complications rates | 30 days
  1. . Incidence of postoperative major complications: The standard for postoperative major complications refers to the short-term complications according to the Clavien-dindo grade, IIIA level and above for serious complications, and when multiple complications occur simultaneously, the highest ranked complication is the subject.
  2. . Postoperative complications are divided into short-term complications after surgery and long-term complications after surgery. (3)Short-term is defined as within 30 days of surgery or the first discharge if the hospital stay is > 30 days.
  (4)Long-term is defined as the period from 30 days or more after the operation or the period between first discharge (the hospital days after surgery >30 days) and 3 years after the operation.
3-year overall survival rate | 36 months
  1. The overall survival is calculated from the day of surgery until death or until the final follow-up date, whichever occurs first.
  2. For survival cases, the end point is the last date that survival was confirmed. If loss to follow-up occurred, the end point is the final date that survival could be confirmed.
3-year recurrence pattern | 36 months
  Definition of recurrence and recurrence date The following situations are regarded as "recurrence"
  1. Recurrence identified by any one image examination (X-ray, ultrasound, computed tomography, magnetic resonance imaging, etc.) and, if there are a variety of imaging examinations, results without contradiction determined "recurrence". The earliest date that the recurrence is found is defined as the "recurrence date".
  2. For cases that lack the use of imaging or a pathological diagnosis, the date of diagnosing the occurrence of clinical recurrence based on clinical history and physical examination is defined as the "recurrence date".
  3. For cases without imaging or clinical diagnosis but with a cytology or tissue biopsy pathological diagnosis of recurrence, the earliest date confirmed by cytology or biopsy pathology is considered the "recurrence date".
  4. A rise in carcinoembryonic antigen or other associated tumor markers alone could not be diagnosed as a relapse.
Overall postoperative morbidity and mortality rates | 30 days
  1. The number of all patients treated with surgery as the denominator and the number of the patients with any intraoperative and postoperative morbidity and mortality as the numerator are used to calculate the proportions.
  2. Postoperative morbidities are divided into short-term and long-term complications after surgery.
  3. Short-term is defined as within 30 days of surgery or the first discharge if the hospital stay is > 30 days.
  4. Long-term is defined as the period from 30 days or more after the operation or the period between first discharge (the hospital days after surgery >30 days) and 3 years after the operation.
  5. Postoperative mortality: patients whose death was identified according to documented intraoperative observation items, including patients who die within 30 days after surgery (including the 30th day) regardless of the causality between death and surgery, and patients who die more than 30 days after surgery.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
Intraoperative tumor rupture rates | 1 day
  Intraoperative tumor rupture rates are used to access the oncological safety of the intervention.
The variation of album | Preoperative 7 days and postoperative 1 and 5 days
  The variation of album in gram/liter on preoperative 7 days and postoperative 1 and 5 days are used to access the postoperative nutritional status and quality of life.
The variation of hemoglobin | Preoperative 7 days and postoperative 1 and 5 days
  The variation of hemoglobin in gram/liter on preoperative 7 days and postoperative 1 and 5 days are used to access the postoperative nutritional status and quality of life.
The variation of white blood cell count | Preoperative 7 days and postoperative 1 and 5 days
  The values of white blood cell count from peripheral blood preoperative 7 days and postoperative 1 and 5 days are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 7 days and postoperative 1 and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood preoperative 7 days and postoperative 1 and 5 days are recorded to access the inflammatory and immune response.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pidhorecky I, Cheney RT, Kraybill WG, Gibbs JF. Gastrointestinal stromal tumors: current diagnosis, biologic behavior, and management. Ann Surg Oncol. 2000 Oct;7(9):705-12. doi: 10.1007/s10434-000-0705-6. PMID 11034250
- [Background] Demetri GD, von Mehren M, Antonescu CR, DeMatteo RP, Ganjoo KN, Maki RG, Pisters PW, Raut CP, Riedel RF, Schuetze S, Sundar HM, Trent JC, Wayne JD. NCCN Task Force report: update on the management of patients with gastrointestinal stromal tumors. J Natl Compr Canc Netw. 2010 Apr;8 Suppl 2(0 2):S1-41; quiz S42-4. doi: 10.6004/jnccn.2010.0116. PMID 20457867
- [Background] Miettinen M, Majidi M, Lasota J. Pathology and diagnostic criteria of gastrointestinal stromal tumors (GISTs): a review. Eur J Cancer. 2002 Sep;38 Suppl 5:S39-51. doi: 10.1016/s0959-8049(02)80602-5. PMID 12528772
- [Background] Karakousis GC, Singer S, Zheng J, Gonen M, Coit D, DeMatteo RP, Strong VE. Laparoscopic versus open gastric resections for primary gastrointestinal stromal tumors (GISTs): a size-matched comparison. Ann Surg Oncol. 2011 Jun;18(6):1599-605. doi: 10.1245/s10434-010-1517-y. Epub 2011 Jan 5. PMID 21207158
- [Background] Melstrom LG, Phillips JD, Bentrem DJ, Wayne JD. Laparoscopic versus open resection of gastric gastrointestinal stromal tumors. Am J Clin Oncol. 2012 Oct;35(5):451-4. doi: 10.1097/COC.0b013e31821954a7. PMID 21552096
- [Background] Koh YX, Chok AY, Zheng HL, Tan CS, Chow PK, Wong WK, Goh BK. A systematic review and meta-analysis comparing laparoscopic versus open gastric resections for gastrointestinal stromal tumors of the stomach. Ann Surg Oncol. 2013 Oct;20(11):3549-60. doi: 10.1245/s10434-013-3051-1. Epub 2013 Jun 21. PMID 23793362
- [Background] Ganai S, Prachand VN, Posner MC, Alverdy JC, Choi E, Hussain M, Waxman I, Patti MG, Roggin KK. Predictors of unsuccessful laparoscopic resection of gastric submucosal neoplasms. J Gastrointest Surg. 2013 Feb;17(2):244-55; discussion 255-6. doi: 10.1007/s11605-012-2095-z. Epub 2012 Dec 8. PMID 23225195
- [Background] De Vogelaere K, Hoorens A, Haentjens P, Delvaux G. Laparoscopic versus open resection of gastrointestinal stromal tumors of the stomach. Surg Endosc. 2013 May;27(5):1546-54. doi: 10.1007/s00464-012-2622-8. Epub 2012 Dec 12. PMID 23233005
- [Background] Bischof DA, Kim Y, Dodson R, Carolina Jimenez M, Behman R, Cocieru A, Blazer DG 3rd, Fisher SB, Squires MH 3rd, Kooby DA, Maithel SK, Groeschl RT, Clark Gamblin T, Bauer TW, Karanicolas PJ, Law C, Quereshy FA, Pawlik TM. Open versus minimally invasive resection of gastric GIST: a multi-institutional analysis of short- and long-term outcomes. Ann Surg Oncol. 2014 Sep;21(9):2941-8. doi: 10.1245/s10434-014-3733-3. Epub 2014 Apr 24. PMID 24763984
- [Background] Lin J, Huang C, Zheng C, Li P, Xie J, Wang J, Lu J. Laparoscopic versus open gastric resection for larger than 5 cm primary gastric gastrointestinal stromal tumors (GIST): a size-matched comparison. Surg Endosc. 2014 Sep;28(9):2577-83. doi: 10.1007/s00464-014-3506-x. Epub 2014 May 23. PMID 24853837
- [Background] Honda M, Hiki N, Nunobe S, Ohashi M, Kiyokawa T, Sano T, Yamaguchi T. Long-term and surgical outcomes of laparoscopic surgery for gastric gastrointestinal stromal tumors. Surg Endosc. 2014 Aug;28(8):2317-22. doi: 10.1007/s00464-014-3459-0. Epub 2014 Feb 25. PMID 24566748
- [Background] Masoni L, Gentili I, Maglio R, Meucci M, D'Ambra G, Di Giulio E, Di Nardo G, Corleto VD. Laparoscopic resection of large gastric GISTs: feasibility and long-term results. Surg Endosc. 2014 Oct;28(10):2905-10. doi: 10.1007/s00464-014-3552-4. Epub 2014 May 31. PMID 24879133
- [Background] Hsiao CY, Yang CY, Lai IR, Chen CN, Lin MT. Laparoscopic resection for large gastric gastrointestinal stromal tumor (GIST): intermediate follow-up results. Surg Endosc. 2015 Apr;29(4):868-73. doi: 10.1007/s00464-014-3742-0. Epub 2014 Jul 23. PMID 25052129
- [Background] Chen K, Zhou YC, Mou YP, Xu XW, Jin WW, Ajoodhea H. Systematic review and meta-analysis of safety and efficacy of laparoscopic resection for gastrointestinal stromal tumors of the stomach. Surg Endosc. 2015 Feb;29(2):355-67. doi: 10.1007/s00464-014-3676-6. Epub 2014 Jul 9. PMID 25005014
- [Background] Dressler JA, Palazzo F, Berger AC, Stake S, Chaudhary A, Chojnacki KA, Rosato EL, Pucci MJ. Long-term functional outcomes of laparoscopic resection for gastric gastrointestinal stromal tumors. Surg Endosc. 2016 Apr;30(4):1592-8. doi: 10.1007/s00464-015-4384-6. Epub 2015 Jul 14. PMID 26169640
- [Background] Nguyen SQ, Divino CM, Wang JL, Dikman SH. Laparoscopic management of gastrointestinal stromal tumors. Surg Endosc. 2006 May;20(5):713-6. doi: 10.1007/s00464-005-0435-8. Epub 2006 Feb 21. PMID 16502196
- [Background] Poskus E, Petrik P, Petrik E, Lipnickas V, Stanaitis J, Strupas K. Surgical management of gastrointestinal stromal tumors: a single center experience. Wideochir Inne Tech Maloinwazyjne. 2014 Mar;9(1):71-82. doi: 10.5114/wiitm.2014.40987. Epub 2014 Feb 26. PMID 24729813
- [Background] Huang CM, Chen QF, Lin JX, Lin M, Zheng CH, Li P, Xie JW, Wang JB, Lu J, Chen QY, Cao LL, Tu RH. Can laparoscopic surgery be applied in gastric gastrointestinal stromal tumors located in unfavorable sites?: A study based on the NCCN guidelines. Medicine (Baltimore). 2017 Apr;96(14):e6535. doi: 10.1097/MD.0000000000006535. PMID 28383420